CLINICAL TRIAL: NCT00925548
Title: A Randomized, Double-blind, Controlled Phase III Study of Stimuvax® (L-BLP25 or BLP25 Liposome Vaccine) in Combination With Hormonal Treatment Versus Hormonal Treatment Alone for First-line Therapy of Post-menopausal Women With Estrogen Receptor (ER)-Positive and/or Progesterone Receptor (PgR)-Positive, Inoperable Locally Advanced, Recurrent, or Metastatic Breast Cancer
Brief Title: STRIDE - STimulating Immune Response In aDvanced brEast Cancer
Acronym: STRIDE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: See termination reason in the below Purpose statement
Sponsor: EMD Serono (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EMR 200038-010; 2008-005544-17 (EudraCT Number)
Record Dates: First submitted 2009-06-17; First posted 2009-06-22 (Estimated); Results first posted 2014-07-24 (Estimated); Last update posted 2014-07-24 (Estimated); Status verified 2014-07

CONDITIONS: Breast Cancer
Keywords: Phase III trial; randomized; cancer vaccine; MUC1; BLP25; advanced breast cancer; postmenopausal breast cancer; immunotherapy of breast cancer; Inoperable locally advanced, recurrent, or metastatic endocrine-sensitive Breast Cancer
MeSH Terms: conditions — Breast Neoplasms; Recurrence | interventions — L-BLP25; Cyclophosphamide; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Investigational Arm (Experimental): Investigational Arm:
  * Pretreatment (Single Dose): 300 milligrams per square meter (mg/m^2) up to a maximum dose of 600 mg of intravenous cyclophosphamide
  * tecemotide (L-BLP25) plus Hormonal Therapy (Standard Dose)
  Interventions: Biological: Tecemotide (L-BLP25) and Hormonal Treatment; Drug: cyclophosphamide
- Control Arm (Active Comparator): Control Arm:
  * Pretreatment (Single Dose): sodium chloride (NaCl) 9 grams per liter (g/L) infusion
  * Placebo plus Hormonal Therapy (Standard Dose)
  Interventions: Biological: Placebo of tecemotide (L-BLP25) and Hormonal Treatment; Drug: sodium chloride (NaCl)

INTERVENTIONS:
Biological: Tecemotide (L-BLP25) and Hormonal Treatment — Investigational Arm:
  Pretreatment (Single Dose) 300 mg/m^2 of intravenous cyclophosphamide in investigational arm to a maximum of 600 milligrams (mg).
  Primary treatment phase:
  Hormonal treatment plus 8 consecutive weekly subcutaneous vaccinations with tecemotide (L-BLP25) 1000 micrograms (actual delivered dose was 930 micrograms)* (Week 1 to 8).
  Maintenance treatment phase:
  Hormonal treatment plus vaccinations with tecemotide (L-BLP25) 1000 micrograms (actual delivered dose was 930 micrograms)* at six-week intervals beginning at Week 14 and continued until Progressive Disease (PD).
  *calculated as mass of lipopeptide (antigen)
  Arms: Investigational Arm
Biological: Placebo of tecemotide (L-BLP25) and Hormonal Treatment — Control Arm:
  Pretreatment (Single Dose) NaCl 9 g/L infusion as a substitute for cyclophosphamide.
  Primary treatment phase:
  Hormonal therapy plus 8 consecutive weekly subcutaneous placebo doses (Week 1 to 8).
  Maintenance treatment phase:
  Hormonal therapy plus placebo doses at six-week intervals beginning at Week 14 and continued until Progressive Disease (PD).
  Arms: Control Arm
Drug: cyclophosphamide — 300 mg/m^2 (to a maximum of 600 mg) of intravenous cyclophosphamide.
  Arms: Investigational Arm
Drug: sodium chloride (NaCl) — NaCl 9 g/L infusion
  Arms: Control Arm

SUMMARY:
EMD Serono has decided to permanently terminate the trial EMR 200038-010 (STRIDE) in the indication of breast cancer following the clinical hold on the investigational new drug application for tecemotide (L-BLP25).

DETAILED DESCRIPTION:
The purpose of the study is to determine whether the addition of the experimental mucinous glycoprotein 1 (MUC1) antigen-specific cancer immunotherapy tecemotide (L-BLP25) to hormonal treatment is effective in prolonging progression-free survival in postmenopausal women with endocrine-sensitive inoperable locally advanced, recurrent or metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women as defined in the protocol
* Estrogen receptor (ER)-positive and/or progesterone receptor (PgR)-positive, histologically or cytologically confirmed primary carcinoma of the breast
* Expressing at least one of the following five human leukocyte antigen (HLA) haplotypes, as centrally assessed by HLA genotyping from whole blood: HLA-A2, -A3, -A11, -B7, or -B35
* Locally advanced, recurrent, or metastatic breast cancer (Subject must have at least one lesion not located in bone)
* Measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST), and inoperable
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Adequate hematologic, hepatic, and renal function within two weeks prior to initiation of therapy, as defined by the protocol
* Other protocol-defined inclusion criteria may apply

Exclusion Criteria:

Disease Status

* PD either during hormonal therapy for early breast cancer (adjuvant therapy) or within 48 months from the initiation of such therapy
* Human epidermal growth factor receptor 2-positive (HER2+) breast cancer as defined in the protocol
* Autoimmune disease that in the opinion of the investigator could compromise the safety of the subject in this study (Exception will be granted for well-controlled Type I diabetes mellitus)
* Recognized immunodeficiency disease, including cellular immunodeficiencies, hypogammaglobulinemia or dysgammaglobulinemia; hereditary or congenital immunodeficiencies
* Past or current history of malignant neoplasm other than breast cancer (BRCA), except for curatively treated non-melanoma skin cancer, in situ carcinoma of the cervix, or other cancer curatively treated and with no evidence of disease for at least five years
* Known active Hepatitis B infection or carrier state and/or Hepatitis C infection, known Human Immunodeficiency Virus infection, or any other infectious process that in the opinion of the investigator could compromise the subject's ability to mount an immune response or could expose her to the likelihood of more and/or severe side effects

Pre-therapies

* Receipt of immunotherapy (for example [e.g.], interferons; tumor necrosis factor; interleukins; growth factors granulocyte macrophage-colony stimulating factor [GM-CSF], granulocyte-colony stimulating factor [G-CSF], macrophage-colony stimulating factor [M-CSF], or monoclonal antibodies), or chemotherapy, within four weeks (28 days) prior to randomization. Note: Subjects who have received monoclonal antibodies for imaging are eligible
* Prior receipt of investigational systemic drugs (including off-label use of approved products) or any kind of systemic treatment (chemotherapy, or immunotherapy), with the exception of hormonal therapy (HT) when given for a period not exceeding 4 weeks (28 days) prior to randomization, for treatment of inoperable, locally advanced, recurrent, or metastatic breast cancer
* Prior radiotherapy to the site of cancer, if only one site will be used for evaluation of tumor response

Prior use of bisphosphonates or concurrent use while on study treatment is allowed

Physiological Function

* Central nervous system disease or brain metastases, as documented by computed tomography (CT) or magnetic resonance imaging (MRI)
* Medical or psychiatric conditions that would interfere with the ability to provide informed consent, communicate side effects, or comply with protocol requirements
* Clinically significant cardiac disease, e.g., cardiac failure of New York Heart Association (NYHA) classes III-IV; uncontrolled angina pectoris, uncontrolled arrhythmia, uncontrolled hypertension, or myocardial infarction in the previous six months, as confirmed by an electrocardiogram (ECG)
* Splenectomy

Standard Criteria

* Need for concurrent treatment with a non-permitted therapy (e.g., concurrent chemotherapy, radiotherapy, systemic immunosuppressive drugs, use of herbal medicines or botanical formulations intended to treat cancer) while on protocol therapy. Palliative radiation to painful bone lesions is allowed
* Participation in another clinical study within 30 days prior to randomization
* Known hypersensitivity to the study drugs
* Known alcohol or drug abuse
* Legal incapacity or limited legal capacity
* Signs and symptoms suggestive of transmissible spongiform encephalopathy, or family members who suffer(ed) from such.
* Subject who could be regarded as "vulnerable" according to International Conference on Harmonisation (ICH) Good Clinical Practice (GCP) guidelines (e.g., the subject's willingness to volunteer in a clinical trial may be unduly influenced by the expectation, whether justified or not, of benefits associated with participation, or of a retaliatory response from senior members of a hierarchy in case of refusal to participate, plus persons kept in detention; persons in nursing homes; subjects in emergency situations; homeless persons; and nomads)
* Any other reason that, in the opinion of the investigator, precludes the subject from participating in this study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2009-09; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Oscar Kashala, MD, PhD, DSc, Study Director — EMD Serono
Locations (29):
- Research Site, Hickory, North Carolina, United States
- Research Site, Bedford Park, SA, Australia
- Austria (2):
  - Research Site, Innsbruck
  - Research Site, Salzburg
- Research Site, Leuven, Belgium
- Czechia (2):
  - Research Site, Pardubice
  - Research Site, Prague
- Germany (10):
  - Research Site, Chemnitz
  - Research Site, Darmstadt
  - Research Site, Frankfurt am Main
  - Research Site, Hamburg
  - Research Site, Kiel
  - Research Site, Lübeck
  - Research Site, München
  - Research Site, Rostock
  - Research Site, Tübingen
  - Research Site, Wiesbaden
- Research Site, Beer Yaakov, Israel
- Research Site, Opole, Poland
- Russia (3):
  - Research Site, Obninsk
  - Research Site, Saint Petersburg
  - Research Site, Tula
- Slovakia (4):
  - Research Site, Bratislava
  - Research Site, Nitra
  - Research Site, Poprad
  - Research Site, Trnava
- Research Site, Johannesburg, South Africa
- South Korea (2):
  - Research Site, Gyeonggi-do
  - Research Site, Seoul

REFERENCES:
- [Derived] Gorodetska I, Samusieva A, Lahuta T, Ponomarova O, Socha O, Kozeretska I. Exploring New Frontiers: Alternative Breast Cancer Treatments Through Glycocalyx Research. Breast J. 2025 May 22;2025:9952727. doi: 10.1155/tbj/9952727. eCollection 2025. PMID 40443562

RESULTS

PARTICIPANT FLOW:
Groups:
- Tecemotide (L-BLP25) + Hormonal Therapy + Cyclophosphamide: Single dose of cyclophosphamide (300 milligrams per square meter [mg/m^2] to a maximum of 600 mg) was administered intravenously, 3 days prior to the start of vaccination, followed by primary treatment phase in which weekly subcutaneous vaccinations with tecemotide (L-BLP25) 1000 micrograms (actual delivered dose was 930 micrograms) along with hormonal treatment were administered for 8 weeks, followed by maintenance treatment phase starting at Week 14 (6 weeks after the last dosing of the primary treatment phase), in which subcutaneous vaccinations with tecemotide (L-BLP25) 1000 micrograms (actual delivered dose was 930 micrograms) along with hormonal treatment were administered every 6 weeks until progressive disease (PD) was documented.
- Placebo + Hormonal Therapy + NaCl 9 g/L: Single dose of sodium chloride (NaCl) 9 grams per liter (g/L) infusion as substitute for cyclophosphamide was administered intravenously, 3 days prior to the start of vaccination, followed by primary treatment phase in which weekly subcutaneous placebo doses matched to tecemotide (L-BLP25) along with hormonal therapy were administered for 8 weeks, followed by maintenance treatment phase starting at Week 14 (6 weeks after the last dosing of the primary treatment phase), in which subcutaneous placebo doses along with hormonal therapy were administered every 6 weeks until progressive disease (PD) was documented.
Period: Overall Study
Arm/Group | Tecemotide (L-BLP25) + Hormonal Therapy + Cyclophosphamide | Placebo + Hormonal Therapy + NaCl 9 g/L
Started | 11 | 5
Completed | 1 | 0
Not Completed | 10 | 5
Not completed — Discontinuation of trial by sponsor | 10 | 5

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received at least one dose of any study treatment (L-BLP25, placebo, cyclophosphamide, saline, or any of the three hormonal therapies).
Groups:
- Placebo + Hormonal Therapy + NaCl 9 g/L: Single dose of sodium chloride (NaCl) 9 g/L infusion as substitute for cyclophosphamide was administered intravenously, 3 days prior to the start of vaccination, followed by primary treatment phase in which weekly subcutaneous placebo doses matched to tecemotide (L-BLP25) along with hormonal therapy were administered for 8 weeks, followed by maintenance treatment phase starting at Week 14 (6 weeks after the last dosing of the primary treatment phase), in which subcutaneous placebo doses along with hormonal therapy were administered every 6 weeks until progressive disease (PD) was documented.
- Total: Total of all reporting groups
Arm/Group | Tecemotide (L-BLP25) + Hormonal Therapy + Cyclophosphamide | Placebo + Hormonal Therapy + NaCl 9 g/L | Total
Number analyzed (Participants) | 11 | 5 | 16
Age, Customized [Number; unit: participants]
  Less than (<) 65 years | 5 | 2 | 7
  Greater than or equal to (>=) 65 years | 6 | 3 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 5 | 16
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS)
Description: PFS was defined as the duration from randomization to first observation of progressive disease (PD) as confirmed by the independent radiological review or death.
Time Frame: Time from randomization to disease progression, death or last tumor assessment, reported between day of first participant randomized i.e. 30 Sep 2009, until end of trial i.e. 27 Aug 2010
Population: Data were not collected as no independent read took place, due to low numbers: the trial was prematurely terminated following the clinical hold on the investigational new drug application for tecemotide (L-BLP25).
Arm/Group | Tecemotide (L-BLP25) + Hormonal Therapy + Cyclophosphamide | Placebo + Hormonal Therapy + NaCl 9 g/L
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Overall Survival (OS) Time
Description: OS time was defined as the time from randomization to death. Participants without event were to be censored at the last date known to be alive or at the clinical cut-off date, whichever was earlier.
Time Frame: Time from randomization to death or last day known to be alive reported between day of first participant randomized i.e. 30 Sep 2009, until end of trial i.e. 27 Aug 2010
Population: Data were not analyzed as the trial was prematurely terminated following the clinical hold on the investigational new drug application for tecemotide (L-BLP25)
Arm/Group | Tecemotide (L-BLP25) + Hormonal Therapy + Cyclophosphamide | Placebo + Hormonal Therapy + NaCl 9 g/L
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Percentage of Participants With Objective Tumor Response
Description: Percentage of participants with objective tumor response was to be reported. An objective response (OR) was defined as a participant having a best overall response of either confirmed complete response (CR) or confirmed partial response (PR) according to Response Evaluation Criteria in Solid Tumors Version 1.0 (RECIST 1.0) as assessed by independent radiological review.
Time Frame: Randomization until the date of first documented progression, until end of trial i.e. 27 Aug 2010
Population: as for outcome 2
Arm/Group | Tecemotide (L-BLP25) + Hormonal Therapy + Cyclophosphamide | Placebo + Hormonal Therapy + NaCl 9 g/L
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Duration of Response
Description: Duration of response is defined as the time from the first assessment of CR or PR until the date of the first occurrence of PD, or until the date of death.
Time Frame: Time from first assessment of CR or PR until PD, death or last tumor assessment, reported between day of first participant randomized i.e. 30 Sep 2009, until end of trial i.e. 27 Aug 2010
Population: as for outcome 2
Arm/Group | Tecemotide (L-BLP25) + Hormonal Therapy + Cyclophosphamide | Placebo + Hormonal Therapy + NaCl 9 g/L
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Percentage of Participants With Clinical Benefit
Description: Clinical Benefit is defined as having achieved at least disease stabilization; that is participants with confirmed CR, PR, or stable disease (SD,) lasting for at least 22 weeks.
Time Frame: Randomization until the date of first documented progression assessed up to end of trial i.e. 27 Aug 2010
Population: as for outcome 2
Arm/Group | Tecemotide (L-BLP25) + Hormonal Therapy + Cyclophosphamide | Placebo + Hormonal Therapy + NaCl 9 g/L
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Time to Progression (TTP)
Description: TTP is defined as the time from date of randomization to the date of radiological diagnosis of PD (censoring for death without progression).
Time Frame: Time from randomization to PD, reported between day of first participant randomized i.e. 30 Sep 2009, until end of trial i.e. 27 Aug 2010
Population: as for outcome 1
Arm/Group | Tecemotide (L-BLP25) + Hormonal Therapy + Cyclophosphamide | Placebo + Hormonal Therapy + NaCl 9 g/L
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Time to Chemotherapy
Description: Time to chemotherapy is defined as the time from date of randomization to the start date of chemotherapy.
Time Frame: Time from randomization to start of chemotherapy, reported between day of first participant randomized i.e. 30 Sep 2009, until end of trial i.e. 27 Aug 2010
Population: as for outcome 2
Arm/Group | Tecemotide (L-BLP25) + Hormonal Therapy + Cyclophosphamide | Placebo + Hormonal Therapy + NaCl 9 g/L
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Functional Assessment of Cancer Therapy-Breast (FACT-B) Questionnaire
Description: FACT-B questionnaire consists of 36 questions; 7 in physical well-being (PWB); 7 in social well-being (SWB); 6 in emotional well-being (EWB); 7 in functional well-being (FWB); 9 in breast cancer subscale (BCS). Trial outcome Index (TOI) was calculated by the sum of the physical well-being (PWB), functional well-being (FWB), and breast cancer scale (BCS) subscales of FACT-B. Total score of subscores or TOI is calculated from each score of question. Higher score means better and lower score means worthier. Score range; 0-28 in PWB; 0-28 in SWB; 0-24 in EWB; 0-28 in FWB; 0-36 in BCS; 0-92 in TOI.
Time Frame: Baseline, Week 9, 20, 32, 44 and end of trial visit
Population: as for outcome 2
Arm/Group | Tecemotide (L-BLP25) + Hormonal Therapy + Cyclophosphamide | Placebo + Hormonal Therapy + NaCl 9 g/L
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: European Questionnaire-5 Dimensions (EQ-5D) Questionnaire
Description: EQ-5D questionnaire is a measure of health status that provides a simple descriptive profile and a single index value. The optional part of the questionnaire was not applied. EQ-5D defines health in terms of mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The 5 items are combined to generate health profiles. These profiles were to be converted to a continuous single index score using a one to one matching. The lowest possible score is -0.59 and the highest is 1.00. Higher scores on the EQ-5D represent a better quality of life (QoL) and lower scores on the EQ-5D represent a worst QoL.
Time Frame: Baseline, Week 9, 20, 32, 44 and end of trial visit
Population: as for outcome 2
Arm/Group | Tecemotide (L-BLP25) + Hormonal Therapy + Cyclophosphamide | Placebo + Hormonal Therapy + NaCl 9 g/L
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Number of Participant Utilizing Healthcare Resources
Description: Healthcare Resource Utilization (HRU) parameters included direct medical resources (e.g., nonscheduled procedures, unplanned hospitalization, outpatient visits), nonmedical resources (e.g., travel, paid and unpaid assistance), and occupational resources (e.g., occupational changes and concerns).
Time Frame: Randomization up to end of trial visit
Population: as for outcome 2
Groups:
- Placebo + Hormonal Therapy + NaCl 9 g/L: Single dose of sodium chloride (NaCl) 9g/L infusion as substitute for cyclophosphamide was administered intravenously, 3 days prior to the start of vaccination, followed by primary treatment phase in which weekly subcutaneous placebo doses matched to tecemotide (L-BLP25) along with hormonal therapy were administered for 8 weeks, followed by maintenance treatment phase starting at Week 14 (6 weeks after the last dosing of the primary treatment phase), in which subcutaneous placebo doses along with hormonal therapy were administered every 6 weeks until progressive disease (PD) was documented.
Arm/Group | Tecemotide (L-BLP25) + Hormonal Therapy + Cyclophosphamide | Placebo + Hormonal Therapy + NaCl 9 g/L
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Serum Carcinoma Antigen (CA) 15-3 Levels
Description: CA 15-3 is a serum marker for breast cancer which is a possible measure for immune response.
Time Frame: Baseline, Week 5, 9, 20, 32, 44 and end of trial visit
Population: as for outcome 2
Arm/Group | Tecemotide (L-BLP25) + Hormonal Therapy + Cyclophosphamide | Placebo + Hormonal Therapy + NaCl 9 g/L
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline (First treatment dose) up to end of trial i.e. 27 Aug 2010
Description: Adverse event (AE): Any untoward medical occurrence/worsening of pre-existing medical condition, whether or not related to study drug.
Arm/Group | Tecemotide (L-BLP25) + Hormonal Therapy + Cyclophosphamide | Placebo + Hormonal Therapy + NaCl 9 g/L
Serious Adverse Events (participants affected / at risk) | 1/11 | 0/5
Other Adverse Events (participants affected / at risk) | 9/11 | 3/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tecemotide (L-BLP25) + Hormonal Therapy + Cyclophosphamide (N=11) | Placebo + Hormonal Therapy + NaCl 9 g/L (N=5)
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tecemotide (L-BLP25) + Hormonal Therapy + Cyclophosphamide (N=11) | Placebo + Hormonal Therapy + NaCl 9 g/L (N=5)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 0
Eye swelling (Eye disorders) | 0 | 1
Ocular hyperaemia (Eye disorders) | 0 | 1
Vision blurred (Eye disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 7 | 1
Vomiting (Gastrointestinal disorders) | 3 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 0
Constipation (Gastrointestinal disorders) | 3 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Eructation (Gastrointestinal disorders) | 1 | 0
Odynophagia (Gastrointestinal disorders) | 1 | 0
Fatigue (General disorders) | 4 | 0
Injection site erythema (General disorders) | 3 | 0
Asthenia (General disorders) | 1 | 1
Injection site haematoma (General disorders) | 0 | 1
Injection site induration (General disorders) | 1 | 0
Injection site pain (General disorders) | 1 | 0
Injection site pruritus (General disorders) | 1 | 0
Injection site swelling (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 0
Nasopharyngitis (Infections and infestations) | 3 | 0
Influenza (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 3 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Dizziness (Nervous system disorders) | 2 | 0
Headache (Nervous system disorders) | 1 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0
Sinus headache (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 1
Depression (Psychiatric disorders) | 1 | 0
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 2 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1
Nail disorder (Skin and subcutaneous tissue disorders) | 1 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 1
Hot flush (Vascular disorders) | 2 | 0
Hypertension (Vascular disorders) | 1 | 0
Jugular vein thrombosis (Vascular disorders) | 1 | 0
Phlebitis (Vascular disorders) | 1 | 0
Thrombophlebitis superficial (Vascular disorders) | 1 | 0
Thrombosis (Vascular disorders) | 0 | 1
Chills (General disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Efficacy data were not analyzed as the trial was prematurely terminated following the clinical hold on the investigational new drug application for tecemotide (L-BLP25)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other